CLINICAL TRIAL: NCT05164211
Title: Didgeridoo Treatment to Improve Pharyngeal Compliance in Obstructive Sleep Apnea-hypopnea Syndrome in Children: Proof-of-concept Study
Brief Title: Didgeridoo Treatment to Improve Pharyngeal Compliance in Obstructive Sleep Apnea-hypopnea Syndrome in Children
Acronym: SASDICO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no inclusion since the opening of the centers (difficulties in recruiting staff which impact the functioning of the services)
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP201130
Record Dates: First submitted 2021-11-19; First posted 2021-12-20 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Didgeridoo
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial, with minimisation criteria, single blind, bicentric
Who Masked: Outcomes Assessor
Masking Description: The nurse performing the rhinopharyngometry measurements does not perform the compliance calculation (primary objective). The measurements from the acoustic pharyngometry are analysed (compliance calculation) by a doctor who does not know the child's randomisation arm. Thus, if the subjects have knowledge of their randomisation group, the assessment of the primary endpoint is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Didgeridoo (Experimental): The children will have 6 didgeridoo lessons given by a teacher spread over 3 months.They will have a didgeridoo at home to practice with.
  Interventions: Other: Didgeridoo
- Absence (No Intervention): The children will have nothing to do.

INTERVENTIONS:
Other: Didgeridoo — the children will have 6 didgeridoo lessons given by a teacher spread over 3 months.
  Arms: Didgeridoo

SUMMARY:
The therapeutic management of Obstructive Sleep Apnoea Syndrome in children remains a debated subject, only otorhinolaryngology surgery (adenoidectomy) has been studied on a large scale. Pathophysiologically, increased pharyngeal collapsibility is a major endotype of the disease and the investigators have shown that this surgery can improve pharyngeal compliance. The development of approaches to treat pharyngeal hypotonia by maxillofacial rehabilitation supports the treatment of this endotype. A study in adults showed a benefit from playing the didgeridoo, a wind instrument, for 3 months, without pathophysiological explanation. The investigators hypothesise that playing this instrument improves pharyngeal compliance (re-education effect) in a similar way to the effect observed after otorhinolaryngology surgery.

This proof-of-concept study aims to demonstrate the effect of didgeridoo in children without syndromic pathology with a formal otorhinolaryngology surgical indication resulting from tonsillar hypertrophy (Brodsky grades III and IV) and symptomatology suggestive of Obstructive Sleep Apnoea Syndrome (Pediatric Sleep Questionnaire score ≥ 0.33). The investigators will take advantage of the long delay in performing the adenoidectomy (~6 months) in their university hospital to evaluate, before the scheduled surgery, the effect of the didgeridoo used for three months.

DETAILED DESCRIPTION:
Randomised controlled trial, with minimisation criteria, single blind, bicentric.

The subjects will be divided into 2 groups, according to the strategy of care before the date of the scheduled surgery: 1. Abstention (routine care) 2. Didgeridoo rehabilitation.

The primary objective is to improve pharyngeal compliance measured non-invasively by acoustic pharyngometry in the didgeridoo arm compared to a no treatment arm.

The secondary objectives are to demonstrate the effect of the didgeridoo on clinical signs associated with Obstructive Sleep Apnoea Syndrome and on an indirect index of apnea-hypopnea during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Clear tonsillar hypertrophy (Brodsky grade III to IV), justifying surgery
* Pediatric Sleep Questionnaire ≥ 0.33
* Discontinuation of any prescribed medication for Obstructive Sleep Apnea Syndrome (anti-histamine and montelukast)
* Access to the Didgeridoo course
* Consent of the holders of parental authority and agreement of the child

Exclusion Criteria:

* Syndromic pathology
* Lack of affiliation to a social security scheme
* Holders of parental authority under guardianship or curatorship

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
pharyngeal compliance | 4 months
  measurement of pharyngeal compliance by acoustic pharyngometry carried out in the sitting and lying position. The associated measurement of the neck circumference (cm) allows the calculation of the pharyngeal compliance in cm3.kPa-1

SECONDARY OUTCOMES:
Quality of the sleep | 4 months
  clinical scores on Pediatric Sleep Questionnaire
Apnea | 4 months
  Apnea Severity Hierarchy score (SHS)
Quality of life | 4 months
  score OSA-18
Desaturation | 4 months
  Desaturation index (IDO3%)
Nocturnal saturation | 4 months
  McGill score
measuring the effect on the surgical indication | 5 months
  number of children for whom the indication for surgery was maintained at the follow-up consultation

CONTACTS AND LOCATIONS:
Overall Officials: Plamen BOKOV, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré; service de Physiologie, Paris, France

IPD SHARING:
Plan to Share IPD: No